CLINICAL TRIAL: NCT06663618
Title: Comparison of Short-term Glucocorticoid Monotherapy and Short-term Glucocorticoid Combined with Mycophenolate Mofetil in the Treatment of IgG4 Related Disease
Brief Title: Short-term Glucocorticoid Combined with MMF for IgG4-RD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wen Zhang (Other)
Responsible Party: Sponsor-Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMF for IgG4-RD
Record Dates: First submitted 2024-10-23; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-09

CONDITIONS: IgG4-related Disease
Keywords: IgG4-related disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — Prednisone; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- short-term glucocorticoid monotherapy (Placebo Comparator): Oral prednison starts at 0.6-0.8mg/kg/d, then tapered and withdrawal in 6 months.
  Interventions: Drug: prednison
- short-term glucocorticoid combined with Mycophenolate mofetil (Experimental): Oral prednison starts at 0.6-0.8mg/kg/d, then tapered and withdrawal in 6 months. Oral Mycophenolate mofetil 0.75g bid for 6 months.
  Interventions: Drug: prednison; Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: prednison — Oral prednison starts at 0.6-0.8mg/kg/d, then tapered and withdrawal in 6 months.
Drug: Mycophenolate mofetil — Oral Mycophenolate mofetil 0.75g bid for 6 months.
  Arms: short-term glucocorticoid combined with Mycophenolate mofetil

SUMMARY:
Comparison of short-term glucocorticoid monotherapy and short-term glucocorticoid combined with MMF in the treatment of IgG4 Related Disease

DETAILED DESCRIPTION:
This is a monocenter, 72-week prospective, randomized controlled study to compare short-term glucocorticoid monotherapy and short-term glucocorticoid combined with MMF in the treatment of IgG4 Related Disease.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old;
2. All patients must meet the comprehensive diagnostic criteria of IgG4-RD revised in Japan in 2020 or the classification criteria of IgG4-RD formulated by ACR/EULAR in 2019;
3. Active IgG4-RD (at least one organ has an IgG4-RD reaction score >=2 at the time of enrollment.)；
4. No previous medication or recurrence after withdrawal.

Exclusion Criteria:

1. Combined with other autoimmune diseases as the main diagnosis.
2. Pregnant or lactating women
3. Patients with malignant tumor
4. Active bacterial, fungal, viral or mycobacterial infections.
5. Severe complications of important organs, and the expected survival time is less than 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
The difference of recurrent rate of IgG4-RD between the two groups | 72 weeks
  Clinical recurrence definition: any item of IgG4-RD Responder Index >=2 points; Recurrence of previously involved organs or involvement of new organs; With or without elevated serum IgG4 levels.

SECONDARY OUTCOMES:
The time of recurrence | 0-72 weeks
  Clinical recurrence definition: any item of IgG4-RD Responder Index >=2 points; Recurrence of previously involved organs or involvement of new organs; With or without elevated serum IgG4 levels.
The changes of IgG4-related disease Responder Index | 72 weeks
  According to international multispecialty validation study of IgG4-related disease Responder Index (November, 2018), Responder Index ≥ 0, and higher scores mean a worse outcome.
The changes of serum IgG4 levels | 72 weeks
  Level of serum IgG4(mg/dL)
The percentages of adverse events | 72 weeks
  Adverse effect of drugs
The changes of PGA | 72 weeks
  Changes of patient global assessment from baseline, score (0-10, higher is worse)
The difference of remission rate of IgG4-RD between the two groups | 72 weeks
  Including complete remission rate, partial remission rate and total response rate.

CONTACTS AND LOCATIONS:
Overall Officials: Wen Zhang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided